CLINICAL TRIAL: NCT03549806
Title: Stanford Cardiac Invasive Electrophysiology Novel Computer Experience (SCIENCE)
Brief Title: Stanford Cardiac Invasive Electrophysiology Novel Computer Experience
Acronym: SCIENCE
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine (CV Medicine), Stanford University
Other Study IDs: SCIENCE
Record Dates: First submitted 2018-04-25; First posted 2018-06-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia; Atrial Flutter; Arrhythmias, Cardiac
Keywords: Atrium, tachyarrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac; Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective Cohort: No study intervention. Patients referred for ablation of atrial arrhythmias will be treated as per operator preference with no study intervention. Data will be collected in de-identified fashion.
  Interventions: Diagnostic Test: No Intervention. Test is computer algorithm.

INTERVENTIONS:
Diagnostic Test: No Intervention. Test is computer algorithm. — Diagnostic algorithms (test) will be run on already acquired clinical data. No study intervention in operator-prescribed clinical ablation. Predictive accuracy of test for study outcome will then be determined in follow-up

SUMMARY:
This study will test the ability of computer algorithms to predict successful ablation therapy for atrial arrhythmias.

DETAILED DESCRIPTION:
Patients will be recruited prospectively from among those undergoing ablation for atrial fibrillation (AF) or atrial tachycardias (AT) which may be reentrant or focal. Each patient will undergo careful data collection, including electrogram data and sites of ablation lesions. Ablation will proceed in operator-dependent fashion, and will not be modified in any way for this study. The research question is whether algorithms based on data such as electrograms and details of the ablation performed can predict which patients will have a successful case. Primary endpoints are measures of clinical success defined by (a) acute termination of atrial arrhythmia during the case; (b) long-term reduction in arrhythmia burden; (c) long-term freedom from arrhythmia. Secondary endpoints include (a) identification of sites of arrhythmia termination; (b) improved clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing catheter ablation for atrial arrhythmias

Exclusion Criteria:

* Inability to sign informed consent
* Expected survival < 1 year
* Extreme comorbidity, such as advanced NYHA Class III/IV heart failure, dialysis, series stroke.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically prescribed ablation for complex atrial arrhythmias will be approached for enrollment. Most are anticipated to be atrial fibrillation or atrial tachyarrhythmias such as post-ablation flutter. Men and women over 21 years and up to 80 years of age will be included.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Reduction in AF burden on follow-up | 2 years
  Reduction in amount of arrhythmia per unit time, compared to prior to the procedure.
Freedom from arrhythmia on follow-up | 2 years
  Absence of arrhythmia, defined by clinical thresholds.

SECONDARY OUTCOMES:
Clinical status as measured by the EQ5D | 2 years
  Patient feeling better subjectively in EQ5D

OTHER OUTCOMES:
Acute Impact of Ablation | Day zero (that is, during procedure).
  Documentation of whether ablation acutely eliminated atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Narayan, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alhusseini M, Vidmar D, Meckler GL, Kowalewski CA, Shenasa F, Wang PJ, Narayan SM, Rappel WJ. Two Independent Mapping Techniques Identify Rotational Activity Patterns at Sites of Local Termination During Persistent Atrial Fibrillation. J Cardiovasc Electrophysiol. 2017 Jun;28(6):615-622. doi: 10.1111/jce.13177. Epub 2017 Mar 20. PMID 28185348
- [Background] Zaman JAB, Sauer WH, Alhusseini MI, Baykaner T, Borne RT, Kowalewski CAB, Busch S, Zei PC, Park S, Viswanathan MN, Wang PJ, Brachmann J, Krummen DE, Miller JM, Rappel WJ, Narayan SM, Peters NS. Identification and Characterization of Sites Where Persistent Atrial Fibrillation Is Terminated by Localized Ablation. Circ Arrhythm Electrophysiol. 2018 Jan;11(1):e005258. doi: 10.1161/CIRCEP.117.005258. PMID 29330332
- [Background] Sahli Costabal F, Zaman JAB, Kuhl E, Narayan SM. Interpreting Activation Mapping of Atrial Fibrillation: A Hybrid Computational/Physiological Study. Ann Biomed Eng. 2018 Feb;46(2):257-269. doi: 10.1007/s10439-017-1969-3. Epub 2017 Dec 6. PMID 29214421
- [Background] Navara R, Leef G, Shenasa F, Kowalewski C, Rogers AJ, Meckler G, Zaman JAB, Baykaner T, Park S, Turakhia MP, Zei P, Viswanathan M, Wang PJ, Narayan SM. Independent mapping methods reveal rotational activation near pulmonary veins where atrial fibrillation terminates before pulmonary vein isolation. J Cardiovasc Electrophysiol. 2018 May;29(5):687-695. doi: 10.1111/jce.13446. Epub 2018 Feb 22. PMID 29377478